CLINICAL TRIAL: NCT01164540
Title: A Randomised, Double-blind, Placebo-controlled, Event Driven, Phase III Study of Rosuvastatin 20 mg Once Daily in the Long Term Prevention of Recurrent Venous Thromboembolism in Patients With Deep Vein Thrombosis or Pulmonary Embolism
Brief Title: Study on the Effect of Rosuvastatin Treatment on the Prevention of Thrombosis in Patients With Previous Thrombosis
Acronym: Du Lac
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to discussion regarding the design of the study.
Sponsor: AstraZeneca (Industry)
Responsible Party: Marketing Company Medical Director, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3560L00093
Record Dates: First submitted 2010-07-08; First posted 2010-07-16 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Venous Thrombosis; Pulmonary Embolism
Keywords: Deep venous thrombosis; Pulmonary embolism; rosuvastatin treatment
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Oral Treatment
  Interventions: Drug: Rosuvastatin (AZD4522)
- 2 (Placebo Comparator): Oral treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosuvastatin (AZD4522) — Oral dose (od) 20 mg
  Other Names: Crestor
  Arms: 1
Drug: Placebo — Oral dose (od)
  Arms: 2

SUMMARY:
This study evaluates whether treatment with rosuvastatin on top of standard anti-coagulant treatment will decrease the risk of recurrent venous thromboembolism and arterial thromboembolic events in patients with previous deep vein thrombosis or pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed Consent.
* Patients with venous thromboembolism who are treated with anti-coagulant according to the current guidelines

Exclusion Criteria:

* Patients in need of or already treated with lipid lowering drugs
* Active liver or kidney disease or dysfunction or muscle disorders
* Unstable medical or psychological condition that interferes with study participation
* Pregnant woman or woman with childbearing potential who are not willing to use contraception
* History of statin-related muscular pain, or hypersensitivity to statins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Any event of venous thromboembolism (i.e. Deep Vein Thrombosis (DVT) and/or fatal or non-fatal Pulmonary Embolism(PE)) | Time to first occurrence in the overall treatment period, with a median treatment period of 9,5 months

SECONDARY OUTCOMES:
All cause mortality | Time to occurrence in the overall treatment period, with a median treatment period of 9,5 months
Any event of the composite of venous thromboembolism or arterial thromboembolism/major adverse cardiovascular event (MACE) | Time to first occurrence in the overall treatment period and during the "on Vitamin K Antagonist (VKA)" treatment period
  Time to first occurrence in the overall treatment period and during the "on (VKA)" treatment period, with an estimated average "on (VKA) treatment period" of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: H. R. Büller, MD, PhD, Principal Investigator — Academic Medical Centre; Michael Cressman, MD, Study Director — AstraZeneca